CLINICAL TRIAL: NCT05932758
Title: Excisional Vacuum-Assisted Breast Biopsy (VAE): Application to Avoid Surgery in Atypical Ductal Hyperplasia and Low/Intermediate Grade Ductal Carcinoma in Situ of the Breast
Brief Title: Excisional Vacuum-Assisted Breast Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Collaborators: Ministero della Salute, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IEO 1856
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Atypical Ductal Hyperplasia; Ductal Carcinoma in Situ
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no excisional biopsy (Other): Patients in this arm underwent to an initial sequence of sampling (less than 4 g of tissue sampled)
  Interventions: Procedure: Not excisional biopsy
- excisional biosy (Experimental): Patients in this arm will undergo a second sequence of biopsy samples (at least 4g sampled)
  Interventions: Procedure: Vacuum-assisted excisional biopsy

INTERVENTIONS:
Procedure: Vacuum-assisted excisional biopsy — at least 4g of tissue sampled (excisional biopsy)
  Arms: excisional biosy
Procedure: Not excisional biopsy — biopsy with less than 4 g of tissue sampled
  Arms: no excisional biopsy

SUMMARY:
The goal of this prospective cohort study is to evaluate the possibility of vacuum-assisted excisional biopsy (VAE) to completely remove the pathology in case of small lesions for Atypical Ductal Hyperplasia (ADH) and low-intermediate grade Ductal Carcinoma in Situ (DCIS).

DETAILED DESCRIPTION:
Surgery is the current standard of care of breast lesions like the Ductal Carcinoma In Situ (DCIS) and the Atypical Ductal Hyperplasia (ADH). However, the survival benefit of surgical resection in patients with such lesions appears to be low, especially for ADH and low-grade DCIS where comorbidity of surgery and prior depression have been reported as important factors related to worse quality of life in these women.

Patients with suspicious breast lesions (BIRADS>3) who are candidates for vacuum assisted breast biopsy will be prospectively select and enroll if the radiological lesion diameter is less than 15 mm.

The investigators will select those patients in whom after an initial sequence of sampling (12 cores), and will check the complete macroscopic removal of the lesion (with radiograms of the biopsied part of the breast). Those patients (complete macroscopic removal, with real-time verification during the procedure) will be randomized into two groups. A first group of patients will finish the biopsy procedure after the first collection sequence (12 cores, 3 grams of tissue taken and complete macroscopic removal). A second group of patients (randomized subdivision) will undergo a second sequence of biopsy samples (other 4 cores and 1 gram of tissue taken) in the same session: the material collected will be sent separately to the pathologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicious breast lesions (BIRADS >3)
* Patients with a lesion <= of 15mm.
* Capable and willing to comply the specific informed consent form
* Patients with ADH biopsy results or low intermediate-grade DCIS
* Patients who will undergo surgery

Exclusion Criteria:

- Patients with psychiatric, addictive, or any disorder, which compromises ability to give informed consent for participation in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with complete removal of lesion | 6 months
  Comparison of the percentage of patients with a lack of pathology (also in situ) at the surgery between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Luca Nicosia, MD, Principal Investigator — European Institute of Oncology IRCCS
Locations (1):
- Breast Imaging Division, Radiology Department, IEO European Institute of Oncology IRCCS, Milan, Italy

REFERENCES:
- [Derived] Nicosia L, Mariano L, Latronico A, Bozzini AC, Bellerba F, Gaeta A, Pesapane F, Mazzarol G, Fusco N, Corso G, Sangalli C, Gialain C, Lazzeroni M, Raimondi S, Cassano E. Exploring non-surgical alternatives for low to intermediate-grade in situ ductal carcinoma of the breast using vacuum-assisted excision: the VACIS protocol. Front Med (Lausanne). 2024 Sep 24;11:1467738. doi: 10.3389/fmed.2024.1467738. eCollection 2024. PMID 39380737